CLINICAL TRIAL: NCT06494657
Title: Frozen Shoulder: A Pragmatic Replicated N-of-1 Case Series Investigating Glucose Levels and Patient Reported Outcomes Following a Corticosteroid Injection.
Brief Title: Frozen Shoulder and Glucose Following Corticosteroid Injection
Status: Not yet recruiting | Type: Observational
Sponsor: Central London Community Healthcare NHS Trust (Other Government)
Collaborators: University of Hertfordshire (Other)
Responsible Party: Sponsor
Other Study IDs: RD24.001
Record Dates: First submitted 2024-07-02; First posted 2024-07-10 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Frozen Shoulder; Adhesive Capsulitis
Keywords: Corticosteroid; Injection; Hyperglycemia
MeSH Terms: conditions — Bursitis; Hyperglycemia | interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Corticosteroid injection — Corticosteroid injection for frozen shoulder

SUMMARY:
The goal of this clinical study is to look at what happens to blood sugar levels in people who have a frozen shoulder, who do not have diabetes after a corticosteroid injection in people with frozen shoulder.

* The primary aim of this study will be to evaluate alterations in glucose levels for people without diabetes, following corticosteroid injection for frozen shoulder.
* The secondary aims are to observe a range of clinical, physiological, and psychosocial outcomes following corticosteroid injection for people with frozen shoulder.

Participants will wear a glucose measuring device, attached to the upper arm collecting readings of glucose levels for 14 days.

Participants will undergo a corticosteroid injection as part of usual care.

DETAILED DESCRIPTION:
Frozen shoulder is regarded one of the most painful conditions to affect the shoulder. It is associated with substantial and prolonged pain that affects sleep and permeates into every aspect of daily function. Epidemiological research suggests the average onset is in the 6th decade, affecting up to 8% of men and 10% of women of working age may be affected. In people with diabetes this figure dramatically increases, with the incidence of frozen shoulder ranging from 10 to 59%.

Injection for frozen shoulder is a well-established treatment option, particularly in the early phase of the condition. The aim of this study is to assess glycaemic changes in a non-diabetic population following a corticosteroid injection. The cardiovascular risk factors associated with developing diabetes, which are increasing globally, because of ageing, smoking, poor diet and lack of physical activity, means there is good reason to understand better the impact of injection for frozen shoulder on the normo-glycaemic population.

A continuous glucose monitor worn on the upper arm, will collect glucose data at multiple timepoints for the 14 days it is worn both before and following the injection. The device is minimally invasive with the use of a small electrochemical sensor inserted under the skin and takes readings of interstitial (between cells, just below the skin).

In the N-of-1 design the 'N' represents a single participant. This design bridges the gap between evidence-based research and clinical care in health conditions. N-of-1 studies are patient centred as participants become more involved in their condition and treatment, setting outcomes due to the close monitoring of participants. When the 'N' is repeated, this may make the findings more generalisable. The CONSORT guidelines for RCTs were extended and the CENT 15 guidelines for N-of-1 trials were developed. A strength of N-of-1 studies as they are focussed on the individual and whilst their comorbidities are stable, they can be included in the study.

For this study, an A-B-A phase design will be used. The initial phase (A) is where repeated glucose measures are automatically obtained via the sensor and uploaded to the website and to check participants glucose levels do not go to the hyper/hypoglycaemic ranges on the day of the injection.

The next phase (B) is the intervention phase where participants will undergo a corticosteroid injection. The final phase (A) is where 'washout' will occur and this will be for the remainder of the life of the sensor. The term 'washout period' refers to ''a period in which no intervention is administered. A washout may be administered between different treatment periods or may act as a period in itself, as in a "reversal" design (to "wash out" the effects of a treatment….'' Glucose data is continually provided by the sensor to the website, which is around 14 days. It will be important to investigate glucose levels for the life of the CGM to assess if any individuals developed hyperglycaemia following the injection.

Day 1 is the day the CGM is attached to the participant. Data will be collected from day 1 but will not be used as part of the analysis as there is less available data collected by the device, resulting in less accurate readings.

Day 2 to day 5, is the pre-injection phase. Day 5 is the day of the injection and up until the point of the injection is included as pre-injection phase. Immediately following the injection is the early phase post injection up to day 8. Day 9 to day 14 is the late phase post injection.

Sampling technique

The process of sample selection will be as follows:

* Potential participants referred to the musculoskeletal physiotherapy department with a diagnosis of primary idiopathic frozen shoulder and fitting the inclusion criteria.
* Purposive sampling technique to include potential participants who may be under-represented, in the health-care setting, particularly if south Asian or black due to the increase incidence of frozen shoulder in these cohorts.
* The sample is derived from the electronic patient record system.

Potential participants will be recruited by their referring GP to the musculoskeletal service. The study aims to have a maximum of 10 completed participant data sets. A literature review of sample size for N-of-1 trials found the average sample size was 13 (range 2 - 428; IQR, 6.5 - 38.5). Other studies had sample sizes of 4 for mobility rehabilitation 8 for virtual reality exercises for neck pain and 4 participants with low back pain and exercise. There is no formal sample size calculation as there are unknown features for example size of the effect. This study is novel and to the best of the chief investigators knowledge there is no other similar study for comparison.

The primary outcome measures are glucose levels pre and post injection and the shoulder pain and disability index (SPADI). A Microsoft Teams channel will enable secure digital data collection and this data will be captured on 2 separate occasions: at baseline and at 3 weeks post-injection. The baseline data will be captured once at the start of participant involvement.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 45 and 65
* Without diabetes or pre-diabetes
* Glenohumeral external rotation range is equally limited actively and passively by at least 50% compared to the contralateral side.

Other glenohumeral movements are equally limited actively and passively compared to the contralateral side in one or more additional planes of movement (such as hand behind the back/shoulder flexion/abduction/scaption).

* The symptoms have been present for at least one month.
* No significant abnormality on plain radiographs.
* Ability to provide informed consent

Exclusion Criteria:

* Aged 44 and under and 66 and over
* People with frozen shoulder secondary to significant shoulder trauma (e.g., dislocation, fracture or full thickness tear requiring surgery) or other causes (e.g., recent breast cancer surgery or radiotherapy)
* People with prediabetes, type 1 and 2 diabetes
* A neurological disease affecting the shoulder
* Evidence of other shoulder disorders (e.g., inflammatory arthritis, rotator cuff disorders, glenohumeral joint instability) or with red flags consistent with the criteria set out by British Elbow and Shoulder Society (Rangan, 2015).
* Primary osteoarthritis of the glenohumeral joint on plain radiograph
* Calcific tendinitis
* Who have received corticosteroid injection for shoulder pain in the last 12 weeks
* On long term steroids or a recent short course of oral steroids
* Currently being treated with coumarin anticoagulants, such as warfarin
* Who have participated in another research study involving an investigational medicinal product in the past 12 weeks
* Significant renal or hepatic impairment
* Any other significant disease which, in the opinion of the Investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study.
* Systemically unwell or with infection
* Pregnant or breastfeeding

Ages: 45 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: People with a Barnet borough GP and with a diagnosis of frozen shoulder
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2024-08-16 (Estimated); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Mean glucose levels | 3 weeks
  The primary biochemical outcome is mean glucose (mmol/dL) levels pre and post injection.
Shoulder Pain and Disability Index | 3 weeks
  The primary clinical outcome is the functional questionnaire 'Shoulder Pain and Disability Index' before and after the injection. The SPADI is a 13-item patient completed instrument. Its categories include "pain" (5 items) and "disability" (8 items), with the total score often described as a percentage, resulting from the summation of each component. Overall total scores range from 0 to 130 with a percentage score of 0 indicating less shoulder disability and 100 indicating more shoulder dysfunction.

SECONDARY OUTCOMES:
Quick Disabilities of the Arm, Shoulder, and Hand | 3 weeks
  The Quick Disabilities of the Arm, Shoulder, and Hand questionnaire is a subset of 11 items from the 30-item Disabilities of the Arm, Shoulder, and Hand and is a self-reported questionnaire in which the response options are presented as 5-point Likert scales. At least 10 of the 11 items must be completed for a score to be calculated and the scores range from 0 (no disability) to 100 (most severe disability). This score was designed be useful in patients with any musculoskeletal disorder of the upper limb.
Pain Self Efficacy Questionnaire | 3 weeks
  The Pain Self Efficacy Questionnaire is a 10-item questionnaire, where patients rate their confidence from 0 points (not at all confident) to 6 points (completely confident). Total scores are calculated by summing the individual items with a range from 0 points (less self-efficacy) to 60 points (more self-efficacy)
Pittsburgh Sleep Quality Index | 3 weeks
  The 19 items are grouped into 7 components, including (1) sleep duration, (2) sleep disturbance, (3) sleep latency, (4) daytime dysfunction due to sleepiness, (5) sleep efficiency, (6) overall sleep quality, and (7) sleep medication use.
  In scoring the Pittsburgh Sleep Quality Index, seven component scores are derived, each scored 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce a global score (range 0 to 21). Higher scores indicate worse sleep quality.
Time in glucose range % | 3 weeks
  The time spent within various glucose ranges pre and post injection

CONTACTS AND LOCATIONS:
Overall Officials: Simon Lewis, Study Chair — Central London Community Healthcare NHS Trustr

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Walker-Bone K, Palmer KT, Reading I, Coggon D, Cooper C. Prevalence and impact of musculoskeletal disorders of the upper limb in the general population. Arthritis Rheum. 2004 Aug 15;51(4):642-51. doi: 10.1002/art.20535. PMID 15334439
- [Background] Wong CK, Levine WN, Deo K, Kesting RS, Mercer EA, Schram GA, Strang BL. Natural history of frozen shoulder: fact or fiction? A systematic review. Physiotherapy. 2017 Mar;103(1):40-47. doi: 10.1016/j.physio.2016.05.009. Epub 2016 Jun 21. PMID 27641499
- [Background] Krasny-Pacini A, Evans J. Single-case experimental designs to assess intervention effectiveness in rehabilitation: A practical guide. Ann Phys Rehabil Med. 2018 May;61(3):164-179. doi: 10.1016/j.rehab.2017.12.002. Epub 2017 Dec 15. PMID 29253607
- [Background] Vohra S, Shamseer L, Sampson M, Bukutu C, Schmid CH, Tate R, Nikles J, Zucker DR, Kravitz R, Guyatt G, Altman DG, Moher D; CENT Group. CONSORT extension for reporting N-of-1 trials (CENT) 2015 Statement. BMJ. 2015 May 14;350:h1738. doi: 10.1136/bmj.h1738. No abstract available. PMID 25976398
- [Background] Shamseer L, Sampson M, Bukutu C, Schmid CH, Nikles J, Tate R, Johnston BC, Zucker D, Shadish WR, Kravitz R, Guyatt G, Altman DG, Moher D, Vohra S; CENT group. CONSORT extension for reporting N-of-1 trials (CENT) 2015: explanation and elaboration. J Clin Epidemiol. 2016 Aug;76:18-46. doi: 10.1016/j.jclinepi.2015.05.018. Epub 2015 Aug 10. PMID 26272791
- [Background] Lobo MA, Moeyaert M, Baraldi Cunha A, Babik I. Single-Case Design, Analysis, and Quality Assessment for Intervention Research. J Neurol Phys Ther. 2017 Jul;41(3):187-197. doi: 10.1097/NPT.0000000000000187. PMID 28628553
- [Background] Punja S, Bukutu C, Shamseer L, Sampson M, Hartling L, Urichuk L, Vohra S. N-of-1 trials are a tapestry of heterogeneity. J Clin Epidemiol. 2016 Aug;76:47-56. doi: 10.1016/j.jclinepi.2016.03.023. Epub 2016 Apr 11. PMID 27079847
- [Background] de la Serna D, Navarro-Ledesma S, Alayon F, Lopez E, Pruimboom L. A Comprehensive View of Frozen Shoulder: A Mystery Syndrome. Front Med (Lausanne). 2021 May 11;8:663703. doi: 10.3389/fmed.2021.663703. eCollection 2021. PMID 34046418
- [Background] Deshmukh H, Wilmot EG, Gregory R, Barnes D, Narendran P, Saunders S, Furlong N, Kamaruddin S, Banatwalla R, Herring R, Kilvert A, Patmore J, Walton C, Ryder REJ, Sathyapalan T. Effect of Flash Glucose Monitoring on Glycemic Control, Hypoglycemia, Diabetes-Related Distress, and Resource Utilization in the Association of British Clinical Diabetologists (ABCD) Nationwide Audit. Diabetes Care. 2020 Sep;43(9):2153-2160. doi: 10.2337/dc20-0738. Epub 2020 Jul 15. PMID 32669277
- [Background] Dyer BP, Rathod-Mistry T, Burton C, van der Windt D, Bucknall M. Diabetes as a risk factor for the onset of frozen shoulder: a systematic review and meta-analysis. BMJ Open. 2023 Jan 4;13(1):e062377. doi: 10.1136/bmjopen-2022-062377. PMID 36599641
- [Background] Kooistra B, Dijkman B, Einhorn TA, Bhandari M. How to design a good case series. J Bone Joint Surg Am. 2009 May;91 Suppl 3:21-6. doi: 10.2106/JBJS.H.01573. PMID 19411496
- [Background] Millar NL, Meakins A, Struyf F, Willmore E, Campbell AL, Kirwan PD, Akbar M, Moore L, Ronquillo JC, Murrell GAC, Rodeo SA. Frozen shoulder. Nat Rev Dis Primers. 2022 Sep 8;8(1):59. doi: 10.1038/s41572-022-00386-2. PMID 36075904